CLINICAL TRIAL: NCT06205173
Title: Explored About Temperature Packing Care to Improve the Quality of Life for Chemotherapy Induced Peripheral Neuropathy (CIPN) in Colorectal Cancer and Gastric Cancer Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201909032RINA
Record Dates: First submitted 2023-11-24; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Gastric Cancer; Chemotherapy-induced Peripheral Neuropathy
Keywords: Hot compressing; Colon Cancer; Colorectal Cancer; Chemotherapy-induced Peripheral Neuropathy; Gastric Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): According to the traditional care model, no interventions are applied to the hands and feet.
- Hot compressing group (Experimental): Temperature control will be maintained within the range of 37-38 degrees Celsius.The application will commence 15 minutes before the administration of Oxaliplatin and conclude 15 minutes after the injection.
  Interventions: Other: Cold compressing
- Cold compressing group (Experimental): Temperature control will be maintained within the range of 12-18 degrees Celsius.The application will commence 15 minutes before the administration of Oxaliplatin and conclude 15 minutes after the injection.
  Interventions: Other: Hot compressing

INTERVENTIONS:
Other: Hot compressing — The intervention in this study will commence 15 minutes before the administration of Oxaliplatin and conclude 15 minutes after the injection. Throughout the process, the patient's local site will be checked every 15 minutes for signs of redness, abnormal sensations, and skin temperature measurement to assess potential harm caused by the applied temperature. If any adverse reactions occur, the intervention will be stopped as necessary.
  Arms: Cold compressing group
Other: Cold compressing — The intervention in this study will commence 15 minutes before the administration of Oxaliplatin and conclude 15 minutes after the injection. Throughout the process, the patient's local site will be checked every 15 minutes for signs of redness, abnormal sensations, and skin temperature measurement to assess potential harm caused by the applied temperature. If any adverse reactions occur, the intervention will be stopped as necessary.
  Arms: Hot compressing group

SUMMARY:
Investigate the effectiveness of cold and hot compress interventions in reducing peripheral neuropathy induced by Oxaliplatin chemotherapy in colorectal cancer and gastric cancer patients. The primary outcome measures include quality of life, and secondary outcome measures encompass the severity of peripheral neuropathy, manual dexterity assessed through finger strength testing, and the effects on microcirculation blood flow in the hands and feet

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect in cancer patients undergoing chemotherapy, with an overall incidence rate of approximately 70-100% for Oxaliplatin. The symptomatology typically manifests as a "glove and stocking" neuropathy, leading to sensory abnormalities that significantly impact patients' activities of daily living and reduce their overall quality of life. Furthermore, it may result in dosage reduction, treatment delays, or interruptions. Studies indicate that residual symptoms persist in 68.1% of patients one month after the completion of chemotherapy, emphasizing the long-term effects of CIPN on post-treatment individuals. Consequently, there is a pressing need for evidence-based preventive intervention research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20 and above, inclusive, can autonomously decide to participate in this study and complete the Participant Consent Form.
* Patients diagnosed with colorectal cancer, receiving chemotherapy for the first time, and being prescribed the standard FOLFOX regimen with Oxaliplatin as the primary agent are eligible. The dosage is 85mg/m2 administered over a 2-hour injection every 14 days, constituting one treatment cycle. A total of 6 treatment cycles will be conducted.

Exclusion Criteria:

* Individuals with an undiagnosed medical condition.
* Individuals with thyroid disorders, diabetes, undergoing dialysis, pregnant, alcohol abusers, and those with immune-related diseases such as lupus erythematosus, scleroderma, dermatomyositis, and rheumatoid arthritis are excluded from the study..
* Individuals with defects in hands, feet, or fingers.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of Cold and Hot Compress Nursing Interventions on the Quality of Life | (1) Before the initiation of the first chemotherapy session. (2) Before the 6th administration of chemotherapy drugs. (3) Before the 12th administration of chemotherapy drugs. (4) Within three months after the completion of the chemotherapy course.
  Quality of Life was measured by EORTC-QLQ-C30.The scale assesses symptoms, functionality, and overall health status/life quality. Each item is transformed to a 0-100 scale according to a standardized scoring procedure.Higher scores indicate more severe symptoms, while in the functionality and overall health status/life quality sections, higher scores signify better conditions.

SECONDARY OUTCOMES:
The effectiveness of Cold and Hot Compress Nursing Interventions on the Quality of Life and severity of Peripheral Neuropathy. | (1) Before the initiation of the first chemotherapy session. (2) Before each administration of chemotherapy drugs (total of 12 times). (3) Within three months after the completion of the chemotherapy course.
  Severity of Peripheral Neuropathy was measured by EORTC QLQ-CIPN2. This assesses symptoms and functional limitations related to sensory, motor, and autonomic nervous system disorders.Each item is transformed to a 0-100 scale according to a standardized scoring procedure.Higher scores indicate more severe symptoms, while in the functionality and overall health status/life quality sections, higher scores signify better conditions.
The effectiveness of Cold and Hot Compress Nursing Interventions on the Severity of Peripheral Neuropathy. | (1) before the initiation of Oxaliplatin treatment, (2)after the completion of the 6th injection until the start of the 7th injection (approximately three months into chemotherapy), (3)Within three months after the completion of the chemotherapy course
  Severity of Peripheral Neuropathy was measured by Total Neuropathy Score-clinical.The assessment includes 3 subjective symptom and 4 objective evaluations, which encompass muscle strength, deep tendon reflexes, vibration threshold, and pinprick sensation. Scores range from 0 (no neuropathy) to 4 (severe neuropathy), higher total score indicating a higher degree of peripheral neuropathy.
The effectiveness of Cold and Hot Compress Nursing Interventions on the Symptoms of Peripheral Neuropathy. | (1) before the initiation of Oxaliplatin treatment, (2)after the completion of the 6th injection until the start of the 7th injection (approximately three months into chemotherapy), (3)Within three months after the completion of the chemotherapy course
  Severity of Peripheral Neuropathy was measured by NCI-CTCAE. Includes evaluations of both motor and sensory nerves. The NCI-CTCAE is primarily based on the severity of adverse events and utilizes a grading system ranging from one (mild) to five (death) to characterize the extent of events. A higher grade indicates more severe symptoms.
The Effectiveness of Cold and Hot Compress Nursing Interventions on the Neurological Changes in the Hands and Feet. | (1) before the initiation of Oxaliplatin treatment, (2)after the completion of the 6th injection until the start of the 7th injection (approximately three months into chemotherapy), (3)Within three months after the completion of the chemotherapy course
  The Effectiveness of Cold and Hot Compress Nursing Interventions on the Neurological Changes in the Hands and Feet through Neuro- electro-physiological study which including upper and lower limb motor nerve conduction measurements, sensory nerve conduction velocity measurements, and F-wave measurements.These were measured by Rehabilitation Physician.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan